CLINICAL TRIAL: NCT05392842
Title: The Potential of Corchorus Olitorius Seeds Buccal Films for Treatment of Recurrent Minor Aphthous Ulcerations in Human Volunteers
Brief Title: Corchorus Olitorius Buccal Films for the Treatment of Recurrent Minor Aphthous Ulcerations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Principal Investigator, Soad Ali, Clinical professor, Deraya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Orafilms
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Aphthous Ulcer Recurrent
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): plain mucoadhesive fast dissolving film
  Interventions: Dietary Supplement: plain mucoadhesive fast dissolving film
- Treated group (Experimental): Corchorus Olitorius Buccal Films
  Interventions: Dietary Supplement: Corchorus Olitorius Buccal fast dissolving Films

INTERVENTIONS:
Dietary Supplement: Corchorus Olitorius Buccal fast dissolving Films — Corchorus Olitorius Buccal fast dissolving Films
  Arms: Treated group
Dietary Supplement: plain mucoadhesive fast dissolving film — plain mucoadhesive fast dissolving film
  Arms: Placebo group

SUMMARY:
A methanol extract of Corchorus olitorius edible plant was perpared for extration of glycosideal compounds. the extract was tested for its efficacy as antiinflammatory and analgesic activity invitro and approved by the biomarkers. a fast dissolvinf mucoadhesive film was prepared by a certain amounts of highly safe polymers for a pilote study on human for treament of Aphthous Ulcerations. two groups of study, placebo and intrvention will be recurited and followed for pain, erthymia and size of ulcers for 6 days.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-65 years old
2. Willingness to participate and sign the informed consent forms
3. Presenting with 1 to 5 aphthous ulcers (less than 72 hours' duration) with a size no greater than 5 mm in diameter
4. An expectation that their ulcers normally take 5 or more days to resolve without treatment

Exclusion Criteria:

* A known history of serious drug hypersensitivities 2. Pregnancy and lactation (Urine hCG-positive) 3. Concurrent clinical conditions that could pose a health risk to the subjects, including serious liver, kidney, and heart dysfunctions 4. A history of an immunologic problem

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
treatment of ulcer | 6 days
  ulcer size by the investigator, the diameter measured as the distance between two oppisit points of the wight area of ulcer

SECONDARY OUTCOMES:
Pain scoring | 6 days
  pain measured by VAS tool, 0 the least pain while 10 the highest one
Erthymia | 6 days
  Erthymia estimated by the dgree of redness by the investgator, the darkest indicadetes the worst one

CONTACTS AND LOCATIONS:
Locations (1):
- Minya university, faculty of medicin, Minya, Minya Governorate, Egypt